CLINICAL TRIAL: NCT05723705
Title: Impact of a European Training Program for Robotic Liver Surgery (LIVEROBOT)
Acronym: LIVEROBOT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: UMC Utrecht (Other); General Hospital Groeninge (Other); Fondazione Poliambulanza Istituto Ospedaliero (Other); Intuitive Surgical (Industry)
Responsible Party: Principal Investigator, Dr. R.J. (Rutger-Jan) Swijnenburg, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: LIVEROBOT; W22_217 # 22.269 (Other: METC Amsterdam UMC)
Record Dates: First submitted 2023-01-25; First posted 2023-02-13 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Liver Diseases; Liver Neoplasm; Liver Cancer; Liver Metastases; Biliary Tract Cancer; Biliary Tract Neoplasms; Biliary Tract Diseases
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; Biliary Tract Neoplasms; Biliary Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: European Multicentre Training Program for Robotic Liver Surgery — LIVEROBOT is a pan-european multicentre training program for robotic liver surgery involving simulation training, a procedure video-library, on and off-site proctoring, and video-assessment.
  Other Names: Robotic Liver Surgery

SUMMARY:
LIVEROBOT is a collaboration of high-volume liver surgical centers in Europe (≥60 liver resections per year), supported by the European-African Hepato-Pancreato-Biliary Association Education Committee (E-AHPBA), and the European Registry of Minimally Invasive Liver Surgery (E-MILS) aiming to support the step-up implementation and safety of advanced surgical expertise of robotic liver surgery (RLS) on a European basis. The LIVEROBOT training program aims to promote the safe implementation of RLS throughout Europe. The data from all patients operated on during a surgeons' participation in the training program will be prospectively gathered allowing for learning curve and outcome analyses.

ELIGIBILITY:
Center/Surgeon Eligibility Criteria:

Prior to admission to the LIVEROBOT training program surgeons must demonstrate laparoscopic experience with a laparoscopic cholecystectomy with OSATS score >3 (reviewed by proctors), participation in the LAELIVE training program or demonstrating more than two-year experience in clinical laparoscopic liver surgery. Additionally, a minimal surgical volume is required for participation. Annual liver surgery volume (open and minimally invasive combined) per two surgeons should be more 60, aiming to reach more than 40 RLS annually. Each participating surgeon should individually perform a minimum of more than 15 hepatectomy procedures annually. Surgeons shall be excluded from the training program if at any point failing to meet the minimal volume criteria (corrected for COVID-19 restrictions).

Inclusion Criteria:

* Age equal or above 18 years
* Eligible for elective minimally invasive and open hepatectomy for malignant, pre-malignant or benign disease located in the liver or biliary tract
* Eligible for both minimally invasive and open surgery according to the operating surgeon
* Fit to undergo the indicated operation according to both the anaesthesiologist and surgeon

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are 18 years or above who are eligible to undergo a robotic hepatectomy for accepted indications.
Sampling Method: Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Textbook Outcome in Liver Surgery (TOLS) | 30 days
  TOLS is a novel composite measure that captures the most desirable surgical outcomes into a single indicator and is defined as the absence of intraoperative incidents of grade ≥ 2 (defined according to the Oslo classification), postoperative bile leakage of grade B or C (according to the severity grading of the International Study Group of Liver Surgery), Clavien-Dindo ≥ Grade 3 complications, 30-day readmission, in-hospital mortality and the presence of R0 resection margin.

SECONDARY OUTCOMES:
CUSUM operative time (Learning curve) | After completion of 50 minor and 50 major robotic liver surgery cases per surgeon
Textbook Outcome in Liver Surgery + (TOLS+) | 30 days
  TOLS+ is an extended definition of TOLS and includes the same variables as TOLS but adds 'prolonged LOS' defined as > 4 days for minor RLS and > 7 days for major RLS.
Performance grading using the modified OSATS score | 2 years (expected)
  As assessed by the proctors through video-review
Conversion to open surgery | at operation completion
Estimated operative blood loss | at operation completion
Blood transfusions | at operation completion
Length of Hospital Stay | Expected 4-10 days depending on if minor or major liver resection
Intra-operative ICG-margin assessment | at operation completion

CONTACTS AND LOCATIONS:
Overall Officials: Rutger-Jan Swijnenburg, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jeroen Hagendoorn, MD PhD, Principal Investigator — UMC Utrecht; Mathieu d'Hondt, MD PhD, Principal Investigator — AZ Groeninge; Mohammed Abu Hilal, MD PhD, Principal Investigator — Poliambulanza Foundation Hospital Brescia

IPD SHARING:
Plan to Share IPD: No